CLINICAL TRIAL: NCT03239821
Title: ANTERO-1: a Clinical Evaluation of an Investigational Device: the VIPUN Balloon Catheter 0.1 Used for the Evaluation of Gastric Motility
Brief Title: Clinical Evaluation of the VIPUN Balloon Catheter 0.1
Acronym: ANTERO-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: S60320
Record Dates: First submitted 2017-07-03; First posted 2017-08-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2017-07

CONDITIONS: Healthy; Motility Disorder; Gastric Emptying
MeSH Terms: interventions — Codeine

STUDY DESIGN:
Intervention Model Description: A single-blinded, monocenter, randomized crossover investigation in healthy volunteers.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo - deflated balloon (Sham Comparator)
  Interventions: Device: VIPUN Balloon Catheter 0.1 deflated; Drug: Placebo
- Placebo - inflated balloon (Placebo Comparator)
  Interventions: Drug: Placebo; Device: VIPUN Balloon Catheter 0.1 inflated
- Codeine - delfated balloon (Active Comparator)
  Interventions: Device: VIPUN Balloon Catheter 0.1 deflated; Drug: Codeine Phosphate
- Codeine - inflated balloon (Active Comparator)
  Interventions: Drug: Codeine Phosphate; Device: VIPUN Balloon Catheter 0.1 inflated

INTERVENTIONS:
Device: VIPUN Balloon Catheter 0.1 deflated — deflation balloon
  Arms: Codeine - delfated balloon; Placebo - deflated balloon
Drug: Codeine Phosphate — 58.8 mg codeïne phosphate
  Arms: Codeine - delfated balloon; Codeine - inflated balloon
Drug: Placebo — Sirupus Simplex
  Arms: Placebo - deflated balloon; Placebo - inflated balloon
Device: VIPUN Balloon Catheter 0.1 inflated — VIPUN Balloon Catheter 0.1 inflated
  Arms: Codeine - inflated balloon; Placebo - inflated balloon

SUMMARY:
The primary aim of this investigation is to assess the safety, feasibility and performance of the VIPUN Balloon Catheter 0.1 in the assessment of gastric motility. The investigation will also assess whether the inflation of the VIPUN Balloon Catheter can stimulate gastric motility and emptying. Furthermore, this investigation will examine whether gastric motility and emptying as measured in this study are correlated.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Aged between and including 18 and 65 years
* BMI between and including 18 and 25
* Understand and able to read Dutch
* In good health on the basis of medical history
* Able to return home without driving a vehicle on visit days 1-4
* Will not operate machines on the same day of treatment (visits 1-4)
* Females subjects of childbearing potential are willing to use adequate contraception
* Refrains from herbal, vitamin and other dietary supplements on the day of the visits

Exclusion Criteria:

Exclusion criteria related to possible influence on end-points:

* Dyspeptic symptoms (assessed with PAGI-SYM questionnaire)
* Using any medication that might affect gastric function or visceral sensitivity
* Known / suspected current use of illicit drugs
* Known psychiatric or neurological illness
* Any gastrointestinal surgery that could influence normal gastric function in the opinion of the investigator

Exclusion criteria related to positioning of the catheter:

* History of heart or vascular diseases like irregular heartbeats, angina or heart attack
* Nasopharyngeal, upper GI or esophageal surgery in the last 30 days
* Suspected basal skull fracture or severe maxillofacial trauma
* History of thermal or chemical injury to upper respiratory tract or esophagus
* Current esophageal or nasopharyngeal obstruction
* Known coagulopathy
* Known esophageal varices

Exclusion criteria related to codeine administration:

* History of opioid dependency
* Known severely decreased kidney or liver function
* Pregnant or breastfeeding women (pregnancy test will be performed on females with childbearing potential)
* Known severe lung disease (e.g. asthma or emphysema)
* Have known side-effects/allergic reactions when taking codeine/morphine
* Known diabetic, fructose intolerance or malabsorption of glucose or galactose or sucrose-isomalase insufficiency.

Exclusion criteria related to Sirupus simplex administration:

• Known diabetic (saccharose), intolerance to or malabsorption of propylene glycol and methyl- and propylparahydroxybenzoate

Exclusion criteria related to nutrients (Fortimel):

• Have a known allergy or intolerance to cow milk, soy, saccharose or any other ingredient of Fortimel Energy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence, frequency, severity, seriousness and relatedness of AEs during the 8 hour visit. | 8 hours
  Incidence, frequency, severity, seriousness and relatedness of AEs
Feasibility: Success rate in completing the procedure (placement and removal VIPUN Balloon Catheter) during the 8 hour visit. | 8 hours
  Success rate in completing the procedure (placement and removal VIPUN Balloon Catheter)
Performance: Motility index (MI) decrease after codeine treatment vs. placebo treatment (inflated balloon) during the 8 hour visit. | 8 hours
  Motility index (MI) decrease after codeine treatment vs. placebo treatment (inflated balloon)

SECONDARY OUTCOMES:
Change in gastric emptying: placebo vs. codeine and deflated vs. inflated balloon | 8 hours
  To explore whether the VIPUN Balloon Catheter 0.1 can influence gastric motility and/or emptying.
Correlation motility index change and gastric emptying time change: placebo vs. codeine (inflated balloon) | 8 hours
  To explore whether there is a correlation between gastric motility and emptying.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven Gasthuisberg, Leuven, Belgium